CLINICAL TRIAL: NCT05873452
Title: Kaitoh Atherectomy System: Peripheral Artery Revascularization of Stenotic/Restenotic Disease Using the Atherectomy System in the Peripheral Arteries
Brief Title: Kaitoh Atherectomy FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIS2021-02
Record Dates: First submitted 2023-03-20; First posted 2023-05-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Kaitoh Atherectomy System (Experimental): Eligible participants will undergo atherectomy using the Kaitoh Atherectomy System.
  Interventions: Device: Kaitoh Atherectomy System

INTERVENTIONS:
Device: Kaitoh Atherectomy System — The Kaitoh Atherectomy System is a handheld device which initiates mechanical rotation of the blade to debulk atherosclerotic lesions.

SUMMARY:
This is a prospective, multi-center and single-arm clinical study to assess the initial safety and effectiveness of the Kaitoh Atherectomy System for the treatment of de novo and/or restenotic lesion(s) in the peripheral arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Rutherford Classification: 3-5 in target limb; Rutherford Classification 3 subjects may be enrolled but will be capped to a limit of 20% of the total enrollment (no more than two Rutherford Class 3 subjects may be enrolled into the study).
* Able and willing to provide informed consent, and comply with follow-up visits at both 30 days and 180 days (6 months)
* Able to comply with antiplatelet therapy as required
* Reference Vessel Diameter is ≥2.0 mm and ≤4.0 mm
* Target lesion length is ≤150 mm
* De novo or restenotic target lesion(s) (except for in-stent restenotic lesion) with stenosis ≥70%, by visual estimation, in a single limb in a single native vessel
* Inflow artery is patent, free from significant lesion stenosis (≥50% stenosis is considered significant) as visually confirmed by angiography. Note: Successful inflow artery treatment is allowed during the index procedure. Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤50% without major vascular complications (absence of flow limiting dissection, embolic event)
* Guidewire has successfully crossed the target lesion(s) within the true lumen

Exclusion Criteria:

* Females who are pregnant or lactating
* Pre-existing illness with life expectancy <1 year
* Known or suspected systemic infection
* Significant gastrointestinal bleeding or any coagulopathy that would preclude the use of anti-platelet therapy
* Subjects with a diagnosis of osteomyelitis and are currently on IV antibiotic therapy
* Endovascular or surgical procedure performed on the target lesion within 3 months of the index procedure
* Subjects who in the opinion of the Investigator have underlying kidney disease and may be at risk for contrast-induced acute kidney injury (AKI)
* Subjects who in the opinion of the Investigator have uncontrolled diabetes
* Allergic to iodine/radiopaque contrast that in the opinion of the Investigator cannot be adequately pre-treated
* History of Coronary Artery Bypass Graft (CABG), unstable angina pectoris, or myocardial infarction within 30 days and/or hemorrhagic stroke within 90 days
* Subjects scheduled to undergo a planned major amputation of the lower limb above the ankle on the target limb
* Allergic to any of the components of the atherectomy device system
* Intraprocedural complications prior to use of the investigational device
* Subjects with a positive COVID-19 test within the last 60 days and/or is symptomatic, at the Investigator's discretion
* Subject with other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre - and post-treatment
* Presence of flow-limiting stenosis (>50% diameter reduction) or occlusion of inflow vessels that was not successfully treated (<50% residual stenosis without flow limiting dissection) before the study intervention/prior to the point of enrollment
* No obvious angiographic evidence of flow to the foot following inflow treatment
* Co-existing aneurysmal disease requiring treatment
* Presence of vessel dissection at the target lesion requiring stent placement
* Clinical/angiographic evidence of distal embolization or acute thrombus
* Severe calcification that is measured >10mm in length and circumferential
* Prior stent placement in the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Freedom from major adverse events (MAEs) | 30 days post-procedure
  Primary Safety
Technical success as confirmed by angiography core lab | through completion of interventional 1 day procedure
  Effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, Principal Investigator — Auckland City Hospital
Locations (2):
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No
Not sharing IPD